CLINICAL TRIAL: NCT05057741
Title: Surgical Prehabilitation of Patients Taken to Major Gastrointestinal Surgery.
Brief Title: Surgical Prehabilitation in Abdominal Surgery
Acronym: SPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Rosario (Other)
Collaborators: Hospital Universitario Mayor Mederi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEI DVO005 1567-CV1324; B- 17-2020 (Other Grant/Funding Number: Centro de Investigaciones Mederi CIMED)
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Older People; Prehabilitation; Surgical Procedure
Keywords: surgical procedure; exercise; nutritional; functional condition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial will be performed. Two study groups will be compared, an experimental group that will receive the educational intervention (multimodal prehabilitation program) and a control group that will continue with the usual management in the Hospital. The project activities will be carried out in Telehealth modality. When the patient accepts to participate in the study and signs the informed consent, he/she will be evaluated by nutrition and physiotherapy. After the initial evaluation that confirms the selection criteria, the patient will be randomly assigned to the study groups, by means of a computer based randomisation program.
  The evaluators of the initial and final conditions of the patients will not know the group to which each patient entering the study has been assigned. The study will be conducted following good clinical practice. The estimated duration of recruitment is sixteen months.
Who Masked: Outcomes Assessor
Masking Description: only the outcome assessor. at the time of reviewing the data and doing the analysis he was blinded to the data. No other form of blinding was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal Prehabilitation (Experimental): Multimodal prehabilitation: exercise, nutrition and relaxation
  Interventions: Behavioral: Multimodal prehabilitation
- Standard of Care (No Intervention): Usual care group: advice of surgeons about self care

INTERVENTIONS:
Behavioral: Multimodal prehabilitation — Patients who will receive a multimodal prehabilitation program consisting of guided self-care activities at home that include exercise, nutrition and relaxation. Information Will be share by e health. Monitored by telephone daily during the first week and three times a week between the second and fourth week.
  The final evaluation of the program will be performed one working day after the control appointment with surgery, which will be scheduled ten days after hospital discharge; and the satisfaction survey will be applied. At 30 days after surgery, a telephone follow-up will be made to inquire about complications and mortality. On that day, self-care recommendations will be given.
  Arms: Multimodal Prehabilitation

SUMMARY:
Randomized clinical trial evaluating changes in functional capacity, postoperative complications and 30-day mortality in patients over 60 years of age undergoing major gastrointestinal surgery who participate in a multimodal prehabilitation program, compared to non-prehabilitated patients.

DETAILED DESCRIPTION:
Introduction: A surgical procedure can have repercussions on the functionality and quality of life of patients, reducing their functional capacity by up to 40%; poor preoperative physical performance increases the risk of perioperative morbidity and mortality by 30% and prolongs functional recovery, increasing the hospital stay of the older adult. Prehabilitation is a preoperative intervention that improves the physical, psychological and nutritional condition of the patient to obtain a better postoperative recovery, mobility and functional independence.

Objective: To evaluate changes in functional capacity, postoperative complications and 30-day mortality in patients over 60 years of age undergoing major gastrointestinal surgery who participate in a multimodal prehabilitation program (exercise, nutrition and relaxation).

Methodology: Randomized clinical trial. Two study groups will be compared, an experimental group that will receive the educational intervention (multimodal prehabilitation program) and a control group that will continue with the usual management in the Hospital. The project activities will be carried out in Telehealth modality due to COVID-19 contagion containment measures.

Expected results: To encourage interprofessional work based on common goals with standardization of data and processes to improve physical condition and reduce post-surgical complications; to establish traceability of care, clinical and functional condition of the patient. It is intended to generate scientific evidence, integrate the research groups Méderi, Rehabilitation Sciences and Clinical Research.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled by the General Surgery, Coloproctology and Hepatobiliary Surgery services
* Cognitive ability to follow instructions,
* Understand the material delivered (basic reading comprehension - through physical or digital media)
* Perform physical exercise.
* Aptitude to exercise according to the cardiovascular risk assessment performed by the treating physician.

Exclusion Criteria:

* Patients scheduled for surgery from the emergency department
* Patients with sepsis,
* Patients with metastatic disease, without curative perspective
* Patients with dysphagia for solid foods
* Patients with incapacitating psychiatric or neurological illnesses
* Patients with documented previous immunosuppression status (corticosteroid users in the 6 weeks prior to the randomisation) and/or HIV
* Diabetic patients, with chronic renal disease, stage 4-5, with renal replacement therapy
* Patients with heart failure decompensated, or that limits the physical exercise
* Patients with dependent mobility
* Patients with history of second primary neoplasm

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
functional capacity | One to six weeks
  Changes in the maximum capacity to carry and use oxygen measured with the 2-minute stationary gait test (2MSG)

SECONDARY OUTCOMES:
postoperative complications | 30 days
  Presence of morbidities, whether or not requiring hospital readmission, generated by the surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Mayor Mederi, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No